CLINICAL TRIAL: NCT01812564
Title: Clinical Utilization of Growth Factors Preparations in the Management of Acute Hamstring Muscle Strain Injury
Brief Title: Use of Platelet Rich Plasma in the Management of Acute Hamstring Muscle Strain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aspetar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GF012
Record Dates: First submitted 2013-02-06; First posted 2013-03-18 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Acute Hamstring Muscle Strain Injury
Keywords: Platelet rich plasma; Interventional; Randomized; Double-blind

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PPP (Placebo Comparator): Placebo: Platelet Poor Plasma
  Under sterile conditions, patients will receive under ultrasound guidance 3 times, 1 cc injection of PPP each, administered by a sports medicine physician (total 3 cc PPP).
  Following the completion of the injections (treatment or control) physiotherapy will commence. Physiotherapy protocols will be based on current ASPETAR best practice models (usual care)
  Interventions: Biological: Platelet Poor Plasma (PPP)
- PRP (Active Comparator): Biological: Platelet Rich Plasma
  Under sterile ultrasound conditions, patients will receive under ultrasound guidance 3 times, 1 cc injection of PRP each, administered by a sports medicine physician (total 3 cc PRP).
  Following the completion of the injections (treatment or control) physiotherapy will commence. Physiotherapy protocols will be based on current ASPETAR best practice models (usual care)
  Interventions: Biological: Platelet Rich Plasma (PRP)
- Physiotherapy (No Intervention): These patients will not receive an injection.
  Following the inclusion physiotherapy will commence. Physiotherapy protocols will be based on current ASPETAR best practice models (usual care)

INTERVENTIONS:
Biological: Platelet Poor Plasma (PPP)
  Arms: PPP
Biological: Platelet Rich Plasma (PRP)
  Arms: PRP

SUMMARY:
The purpose of this study is to evaluate the therapeutic benefit of utilizing complex growth factor preparations (Platelet Rich Plasma (PRP) in the management of acute hamstring injuries.

The hypothesis is that the time to return to sport is shorter in the patient group treated with Complex Growth Factor Preparations (PRP) in combination with exercise therapy in comparison with 2 control groups:

* the patient group treated with Platelet Poor Plasma (PPP) injections in combination with exercise therapy (control injection AND usual care).
* the patient group treated with exercise therapy (usual care)

ELIGIBILITY:
Inclusion Criteria:

* Acute onset posterior thigh pain
* MRI confirmed Grade I, II hamstring lesions
* < 5 days from injury
* Able to perform Physiotherapy at ASPETAR (5 sessions/week)
* Available for follow-up
* Male
* Age > 18 years

Exclusion Criteria:

* Diabetes, immuno-compromised state
* Overlying skin infection
* Re-injury or Chronic ongoing hamstring injury
* Unwilling to comply with follow up
* Contraindication to MRI
* Needle Phobia
* Bleeding disorder or other medical contraindication to injection
* Medication increasing bleeding risk (e.g. Plavix)
* Concurrent other injury inhibiting rehabilitation

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time to Return to Play | Patients will be followed for the duration of time to return to play with an expected average of 27 days and up to 1 year.
  Time to return to full sports activity; either training or match play.

SECONDARY OUTCOMES:
Recurrent hamstring lesions. | 2 months after return to play, 1 year after return to play.

OTHER OUTCOMES:
Pain during walking, jogging, running, sprinting, acceleration and during training. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
Pain with isometric contraction against resistance assessed with the visual analogue scale(VAS). | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
Length and width of pain area during palpation and location of pain on palpation. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
Passive straight leg raising test. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
Full knee extension test at rest. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
90 degrees hip flexion test. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
(Painful) resisted knee flexion test at 90 degrees. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
Pain with resisted hip extension test at 30 degrees. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
Slump test. | Once every 7 days from the inclusion date until the time to return to play. (The expected average return to play time is 27 days)
MRI scoring. | 3 weeks after date of injury.
Hamstring strength | At time of return to play (The expected average return to play time is 27 days)
Adverse effects. | Once every 7 days from the inclusion date until the time to return to play (the expected average return to play time is 27 days), 2 months after return to play, at the end of the sport season, and at 1 year after return to play.

CONTACTS AND LOCATIONS:
Overall Officials: Hakim Chalabi, MD, Study Director — Aspetar; Bruce Hamilton, MD, Principal Investigator — Aspetar
Locations (1):
- Aspetar; Qatar Orthopaedic and Sports Medicine Hospital, Doha, Qatar

REFERENCES:
- [Background] Ekstrand J, Healy JC, Walden M, Lee JC, English B, Hagglund M. Hamstring muscle injuries in professional football: the correlation of MRI findings with return to play. Br J Sports Med. 2012 Feb;46(2):112-7. doi: 10.1136/bjsports-2011-090155. Epub 2011 Dec 5. PMID 22144005
- [Background] de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. Platelet-rich plasma injection for chronic Achilles tendinopathy: a randomized controlled trial. JAMA. 2010 Jan 13;303(2):144-9. doi: 10.1001/jama.2009.1986. PMID 20068208
- [Background] Hamilton BH, Best TM. Platelet-enriched plasma and muscle strain injuries: challenges imposed by the burden of proof. Clin J Sport Med. 2011 Jan;21(1):31-6. doi: 10.1097/JSM.0b013e318205a658. PMID 21200168
- [Background] Hamilton B, Knez W, Eirale C, Chalabi H. Platelet enriched plasma for acute muscle injury. Acta Orthop Belg. 2010 Aug;76(4):443-8. PMID 20973348
- [Derived] Zein MI, Mokkenstorm MJK, Cardinale M, Holtzhausen L, Whiteley R, Moen MH, Reurink G, Tol JL; Qatari and Dutch Hamstring Study Group. Baseline clinical and MRI risk factors for hamstring reinjury showing the value of performing baseline MRI and delaying return to play: a multicentre, prospective cohort of 330 acute hamstring injuries. Br J Sports Med. 2024 Jul 1;58(14):766-776. doi: 10.1136/bjsports-2023-107878. PMID 38729628
- [Derived] Whiteley R, van Dyk N, Wangensteen A, Hansen C. Clinical implications from daily physiotherapy examination of 131 acute hamstring injuries and their association with running speed and rehabilitation progression. Br J Sports Med. 2018 Mar;52(5):303-310. doi: 10.1136/bjsports-2017-097616. Epub 2017 Oct 30. PMID 29084725
- [Derived] Jacobsen P, Witvrouw E, Muxart P, Tol JL, Whiteley R. A combination of initial and follow-up physiotherapist examination predicts physician-determined time to return to play after hamstring injury, with no added value of MRI. Br J Sports Med. 2016 Apr;50(7):431-9. doi: 10.1136/bjsports-2015-095073. Epub 2016 Feb 3. PMID 26843538
- [Derived] Wangensteen A, Almusa E, Boukarroum S, Farooq A, Hamilton B, Whiteley R, Bahr R, Tol JL. MRI does not add value over and above patient history and clinical examination in predicting time to return to sport after acute hamstring injuries: a prospective cohort of 180 male athletes. Br J Sports Med. 2015 Dec;49(24):1579-87. doi: 10.1136/bjsports-2015-094892. Epub 2015 Aug 24. PMID 26305004
- [Derived] Hamilton B, Tol JL, Almusa E, Boukarroum S, Eirale C, Farooq A, Whiteley R, Chalabi H. Platelet-rich plasma does not enhance return to play in hamstring injuries: a randomised controlled trial. Br J Sports Med. 2015 Jul;49(14):943-50. doi: 10.1136/bjsports-2015-094603. PMID 26136179
- [Derived] De Vos RJ, Reurink G, Goudswaard GJ, Moen MH, Weir A, Tol JL. Clinical findings just after return to play predict hamstring re-injury, but baseline MRI findings do not. Br J Sports Med. 2014 Sep;48(18):1377-84. doi: 10.1136/bjsports-2014-093737. Epub 2014 Jul 18. PMID 25037201